CLINICAL TRIAL: NCT00969358
Title: Evaluation of a Rehabilitation Program After Lung Surgery (Prospective Observational Study)
Brief Title: Evaluation of a Rehabilitation Program After Lung Surgery
Status: Completed | Type: Observational
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/12
Record Dates: First submitted 2009-08-28; First posted 2009-09-01 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Thoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Fast track programs, multimodal therapy strategies, have been introduced in many surgical fields to minimize postoperative morbidity and mortality. This study is intended to evaluate a rehabilitation program in comparison with a historical series.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* ASA 1, 2 or 3
* lung surgery (postero-lateral or axillary approach)
* epidural analgesia

Exclusion Criteria:

* preoperative oxygen therapy
* lack of autonomy
* unstable coronary artery disease
* FEV1 < 50%
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
length of postoperative hospital stay | end of hospitalisation

SECONDARY OUTCOMES:
Program Monitoring | end of hospitalisation
postoperative complications | end of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (1):
- Dept of Anesthesiology, Hôpital Foch, Suresnes, France